CLINICAL TRIAL: NCT00693654
Title: A Controlled Comparative Study of the Efficacy of SARNA Sensitive Lotion for Treatment of Uremic Pruritus in Adult Hemodialysis Patients
Brief Title: Comparative Study of the Efficacy of SARNA Sensitive Lotion for Treatment of Uremic Itch in Adult Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: Stiefel, a GSK Company (Industry)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00000656; 31648 (Other: WakeForest)
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Pruritis
Keywords: Uremic Pruritis
MeSH Terms: conditions — Pruritus | interventions — mRNA Vaccines; cetyl alcohol, propylene glycol, sodium lauryl sulfate non-lipid cleansing lotion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sarna Lotion (Experimental): 1% pramoxine Sarna lotion
  Interventions: Drug: Sarna
- Placebo Cetaphil lotion (Placebo Comparator): Placebo Cetaphil lotion
  Interventions: Drug: Cetaphil

INTERVENTIONS:
Drug: Sarna — Active Ingredient: Pramoxine Hydrochloride Inactive ingredients:Benzyl Alcohol, Carbomer 940, Cetyl Alcohol, Dimethicone, Glyceryl Stearate (&) PEG-100 Stearate, Isopropyl Myristate, Petrolatum, PEG 8 Stearate, Purified Water, Stearic Acid, Sodium Hydroxide
  Arms: Sarna Lotion
Drug: Cetaphil — Purified Water, Glycerin, Hydrogenated Polyisobutene, Cetearyl Alcohol, Ceteareth 20, Macadamia Nut Oil, Dimethicone, Tocopheryl Acetate, Stearoxytrimethylsilane, Stearyl Alcohol, Panthenol, Farnesol, Benzyl Alcohol, Phenoxyethanol, Acrylates/C10-30 Alkyl Acrylate Crosspolymer, Sodium Hydroxide, Citric Acid
  Other Names: Cetaphil Lotion
  Arms: Placebo Cetaphil lotion

SUMMARY:
The purpose of this research study is to evaluate the efficacy of SARNA Sensitive Lotion in the treatment of uremic pruritus in adult hemodialysis patients in a double-blind Controlled comparative trial.

DETAILED DESCRIPTION:
This was a 4-week, randomized, double-blind, controlled study. Fourteen subjects received treatment lotion (1% pramoxine HCl) and the remaining 14 received a bland emollient (Cetaphil lotion). A target lesion limited to one anatomic site, excluding face and genitals, was selected at baseline. Each subject was instructed to apply lotion twice daily to all affected areas of pruritus for four weeks. The use of any other topical or systemic medication to treat uremic pruritus was not permitted while participating in the study. Subjects were clinically evaluated for erythema, xerosis, lichenification and overall severity at baseline, week 1, and week 4 (end of study)

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years of age to 70 years of age.
* A diagnosis of moderate to severe pruritus.
* At least 3 episodes of itch over a period of 2 weeks, each lasting for 2 minutes or more.
* Symptoms of itch in regular pattern over 6 months.
* Itch Visual analog scale (VAS) of 3cm or more out of 10 cm.
* All subjects will be end stage renal failure patients undergoing hemodialysis for at least 3 months, who have substantial pruritus for more than 6 months. Substantial pruritus is defined as persistent pruritus impairing sleep or daytime activity.
* Ability and willingness to follow all study procedures, attend all scheduled visits, and successfully complete the study
* The ability to understand and sign a written informed consent form, which must be obtained prior to treatment.

Exclusion Criteria:

* Presence of infection (as defined by the investigator) on the area to be treated.
* Subjects with history of pruritus predating renal failure and subjects with skin disease unrelated to uremia, such as atopic dermatitis, will be excluded.
* Use of systemic medications for treatment of pruritus including corticosteroids within the past 4 weeks and during the study.
* Use of topical medications for treatment of pruritus, including corticosteroids, within the past week.
* Pregnant women, women who are breast feeding, or women of child bearing potential who are not practicing an acceptable method of birth control (abstinence, birth control pill/patch, barrier with spermicidal jelly, IUD, etc.), as determined by the investigator. Acceptable contraception must be used during the entire study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-11; Primary Completion 2006-11 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Fleischer, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 11/6/06 to 11/27/06 from the Salem Kidney Center in Winston Salem, NC.
Pre-assignment Details: Subjects were randomized so that half received Sarna lotion to be applied twice daily to all areas of pruritus, the other half applied placebo lotion twice daily to areas of pruritus.
Groups:
- Pramoxine Lotion: Active Medicated Pramoxine Lotion (Sarna) applied topically twice daily to areas of pruritus
- Placebo Cetaphil Lotion: Placebo lotion (Cetaphil) applied twice daily to areas of pruritus
Period: Overall Study
Arm/Group | Pramoxine Lotion | Placebo Cetaphil Lotion
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active: Active Medicated Lotion (Sarna)
- Placebo: Placebo lotion (Cetaphil)
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (13.6) | 58.0 (7.54) | 53.5 (7.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Investigator Global Assessment
Description: Investigator's Global Assessment Disease Severity is based on the following scale:
  0 = completely clear: except for possible residual hyper pigmentation
  1. = almost clear: very significant clearance (about 90%)
  2. = Marked improvement: significant improvement (about 75%)
  3. = Moderate improvement: intermediate between slight and marked; representing about 50% improvements
  4. = Slight improvement: some improvement (about 25%); however, significant disease remaining
  5. = No change (moderate to severe disease)
  6. = Worse
Time Frame: Disease severity assessed at baseline and 4 weeks, week 4 reported
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Active: Active Medicated Pramoxine Lotion (Sarna)
Arm/Group | Active | Placebo
Number analyzed (Participants) | 14 | 14
units on a scale | 2.63 (0.37) | 2.32 (0.36)

2. Secondary Outcome: VAS of Pruritus
Description: Subject's self assessment of itching based on a 100 mm visual analog scale with 0 being no itching and 10 being most severe itching
Time Frame: Assessed at baseline and 4 weeks, week 4 reported
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 14 | 14
units on a scale | 2.73 (0.12) | 2.82 (0.12)

ADVERSE EVENTS:
Arm/Group | Active | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No